CLINICAL TRIAL: NCT02083159
Title: C1q/TNF-related Proteins in Non-Alcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: NAFLD(CTRP)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with NAFLD

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is characterized by an accumulation of fat in the liver, which is one of the most common forms of chronic liver disease in developed countries. In western countries, the prevalence of NAFLD in the general population is estimated to be 20-30%; in obese populations, this increases to 57.5-74%. But, it hasn't been clearly elucidated yet regarding the underlying disease pathophysiology and treatmet strategy.

Recently, members of the C1q/tumor necrosis factor-related protein (CTRP) family have been reported to share structural homology with adiponectin. To date, 15 CTRP family members have been found that might play major roles in glucose metabolism and inflammation.

The investigators tried to clarify the relationship between CTRP family and NAFLD in Korean men and women.

ELIGIBILITY:
Inclusion Criteria:

* 20<age<80
* apparently healthy subjects

Exclusion Criteria:

* a history of CVD
* diabetes
* stage 2 hypertension
* malignancy
* severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects who visited for a routine health check-up at the Health Promotion Center of Korea University Guro Hospital were enrolled using predefined inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
serum concentration of CTRP-1, 3, or 9 in the subjects with/without NAFLD | at enrollment

SECONDARY OUTCOMES:
The relationships of serum CTRPs/adiponectin levels with cardiometabolic risk profiles | at enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Univ. Guro Hospital, Seoul, South Korea